CLINICAL TRIAL: NCT07163312
Title: Prospective Observational Cohort Study of Knee Pain and Function After Endovenous Treatment for Lower Limb Varicose Veins
Brief Title: Knee Pain Relief After Endovenous Treatment for Lower Limb Varicose Veins: A Prospective Observational Study
Acronym: VV-KNEE
Status: Not yet recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Ph.D , Chief Physician of Vascular Surgery , Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Other Study IDs: chengduUTCM knee
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Varicose Veins of Lower Limb; Chronic Venous Insufficiency, CVI; Knee Pain Chronic; Knee Osteoarthritis
MeSH Terms: conditions — Blindness, Cortical; Osteoarthritis, Knee | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovenous Ablation for Varicose Veins — Participants will receive standard endovenous treatment for lower limb varicose veins as part of their routine clinical care. The procedure may include radiofrequency ablation (RFA), endovenous laser ablation (EVLA), or other accepted thermal ablation techniques, with or without adjunctive phlebectomy or foam sclerotherapy if clinically indicated. The intervention is performed under tumescent local anesthesia by vascular surgeons according to established guidelines. No experimental techniques or investigational devices are used.
  Other Names: Endovenous Thermal Ablation (Radiofrequency Ablation or Endovenous Laser Ablation); Endovenous Treatment for Varicose Veins; Standard Varicose Vein Surgery

SUMMARY:
This study will observe patients with lower limb varicose veins who also have knee pain. Many patients with varicose veins experience swelling, heaviness, or aching in the legs, and some also report pain in or around the knee. Previous studies suggest that venous reflux and poor circulation may increase discomfort in the knee, especially when knee osteoarthritis is present.

The purpose of this study is to evaluate whether treatment of varicose veins with standard endovenous procedures can improve knee pain and function. Participants will undergo standard vein treatment as part of their clinical care. We will follow them for changes in knee pain, quality of life, and leg symptoms over time.

This study does not assign patients to experimental interventions. Instead, it collects information before and after treatment to better understand the relationship between varicose veins and knee pain relief. Findings from this study may help doctors identify which patients are most likely to benefit from venous treatment in terms of both leg and knee symptoms.

ELIGIBILITY:
Inclusion Criteria:

Adults aged ≥18 years. Clinical diagnosis of lower limb varicose veins with documented venous reflux on duplex ultrasound (CEAP C2-C4).

Presence of knee pain lasting ≥4 weeks prior to enrollment, confirmed by patient-reported VAS/NRS ≥3 at baseline.

Planned to undergo standard endovenous treatment (radiofrequency ablation, endovenous laser ablation, or equivalent).

Ability to provide informed consent and complete study questionnaires.

Exclusion Criteria:

Prior surgery or endovenous ablation for varicose veins in the same limb. History of inflammatory arthritis (e.g., rheumatoid arthritis, gout) or other systemic rheumatologic disease.

Recent acute knee injury (ligament, meniscus, fracture) within 6 months. Prior knee replacement or major knee surgery. Recent intra-articular injection or arthroscopy (<3 months). Known deep vein thrombosis or history of pulmonary embolism within the past 6 months.

Severe peripheral arterial disease (ABI <0.8). Pregnancy or breastfeeding. Inability to comply with follow-up schedule or complete questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients with clinically significant lower limb varicose veins (CEAP C2-C4) who also report knee pain. Participants are recruited from vascular surgery outpatient clinics and will undergo standard endovenous treatment as part of their clinical care. The study will observe changes in knee pain, function, and venous symptoms before and after treatment. Patients with advanced joint disease, systemic inflammatory disorders, or recent knee surgery are excluded to minimize confounding factors.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Score (VAS) | From baseline to 3 months after treatment
  Visual Analog Scale (VAS, 0-10 cm)

SECONDARY OUTCOMES:
Change in Knee Function and Symptoms | Baseline, 1 month, 3 months, and 6 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) evaluates knee-related pain, stiffness, and functional limitations.Scoring Range: 0 to 96, with higher scores indicating worse symptoms and greater functional impairment.
Change in Venous Clinical Severity Score (VCSS) | Baseline, 1 month, 3 months, and 6 months.
  The Venous Clinical Severity Score (VCSS) assesses the severity of chronic venous disease and varicose vein-related symptoms.Scoring Range: 0 to 30, with higher scores indicating more severe venous disease.
Change in Aberdeen Varicose Vein Questionnaire (AVVQ) | Baseline, 1 month, 3 months, and 6 months.
  The Aberdeen Varicose Vein Questionnaire (AVVQ) measures varicose vein-specific quality of life.Scoring Range: 0 to 100, with higher scores indicating worse quality of life.
Change in Health-Related Quality of Life | Baseline, 1 month, 3 months, and 6 months
  The Chronic Venous Insufficiency Questionnaire (CIVIQ-14) is a 14-item disease-specific instrument used to assess quality of life in patients with chronic venous disease. It covers domains of pain, physical function, and psychological impact. Scoring Range: 0 to 100, with higher scores indicating worse quality of life.
Use of Analgesic Medications | 6 months.
  Number of patients using NSAIDs or other pain medications for knee pain.
Adverse Events Related to Procedure | Within 6 months after procedure.
  Number and type of adverse events (nerve injury, phlebitis, DVT, infection).

IPD SHARING:
Plan to Share IPD: No
Plan Description: Individual participant data (IPD) will not be shared because the study is observational, single-center, and involves limited sample size. Data will be used only for the purpose of this research project and protected according to institutional regulations.

REFERENCES:
- [Background] Lesnyak OM, Zubareva EV, Goncharova MG, Maksimov DM. [Lower extremity venous diseases in primary knee osteoarthritis]. Ter Arkh. 2017;89(5):53-59. doi: 10.17116/terarkh201789553-59. Russian. PMID 28631699
- [Background] Zhang X, Joy DC. A simple specimen holder for EBIC imaging on the Hitachi S800. Microsc Res Tech. 1993 Oct 1;26(2):182-3. doi: 10.1002/jemt.1070260214. No abstract available. PMID 8241555
- [Background] Reading AE, Everitt BS, Sledmere CM. The McGill Pain Questionnaire: a replication of its construction. Br J Clin Psychol. 1982 Nov;21 (Pt 4):339-49. doi: 10.1111/j.2044-8260.1982.tb00571.x. PMID 7171883